CLINICAL TRIAL: NCT05129150
Title: Cognitive Disorders and Brain Pulse
Acronym: COG-PULCE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI21-COG PULCE
Record Dates: First submitted 2021-10-12; First posted 2021-11-22 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Neurocognitive Disorders
Keywords: Brain pulse; ultrasound
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- assessment of cognitive functions: Assessment of cognitive disorders with an ultrasound examination performed in routine care during a day hospital.
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Ultrasound examination with Tissue Pulsatility Imaging (TPI) TPI is a relatively simple, rapid and non-invasive ultrasound examination which consists of applying a standard ultrasound probe to the acoustic window of the temporal bone to first measure the velocity of the middle cerebral artery in Doppler mode and secondly the cerebral pulsatility (CP) of a region of approximately 10cm2 centred on the middle cerebral artery in B-Echo mode. After collecting the information, the TPI examination will be performed by MRRC staff specially trained in TPI by engineers. The duration of the examination is between 20 and 30 minutes, including hardware installation. Four 30-second PC acquisitions will be collected per examination, with the patient lying supine on the bed in the day hospital room, then one measurement every minute for 3 minutes after standing.

SUMMARY:
Following an initial consultation with a memory, resources and research centre (MRRC) doctor, a day hospital may be prescribed to carry out an assessment of cognitive disorders. Patients are then usually followed up in consultation at least once a year, in the framework of a new day hospital and/or consultations with a MRRC doctor.

DETAILED DESCRIPTION:
Patients will be included at the time of the day hospital assessment. All patients received in the day hospital of the MRRC of Tours will be offered the TPI examination. The patients included will be followed up for a period of 5 years and the TPI examination will be repeated according to the same modalities, as part of their follow-up at the MRRC and/or in the context of a new day hospital if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient benefiting from a day hospital at the MRRC of the CHU of Tours for assessment of cognitive functions

Exclusion Criteria:

* Refusal of TPI ultrasound examination
* Patients who opposed to data processing
* Patients under judicial protection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient benefiting from a day hospital at the MRRC of the CHU of Tours for assessment of cognitive functions
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
maximum amplitude of brain movements | one a year from inclusion visit to 5 years
  Measurement by ultrasound between patients with Minor Neurocognitive Disorders (mNCD) and Major Neurocognitive Disorders (MNCD).
mean of brain movements | one a year from inclusion visit to 5 years
  Measurement by ultrasound between patients with Minor Neurocognitive Disorders (mNCD) and Major Neurocognitive Disorders (MNCD).
standard deviation of brain movements | one a year from inclusion visit to 5 years
  Measurement by ultrasound between patients with Minor Neurocognitive Disorders (mNCD) and Major Neurocognitive Disorders (MNCD).
powers in frequency analysis | one a year from inclusion visit to 5 years
  Measurement by ultrasound between patients with Minor Neurocognitive Disorders (mNCD) and Major Neurocognitive Disorders (MNCD).

SECONDARY OUTCOMES:
Brain pulse | one a year from inclusion visit to 5 years
  Longitudinal comparison between converter patients (patients with mNCD progressing to MNCD) and non-converters patients
Brain pulse | one a year from inclusion visit to 5 years
  Cross-sectional and longitudinal analysis between the different types of pathologies underlying NCD (Alzheimer's disease, Vascular NCD, Frontotemporal Lobar Degeneration, Lewy body disease, etc.) according to the Diagnostic and Statistical Manual of mental disorders criteria for these pathologies
Hippocampal volume | one a year from inclusion visit to 5 years
  Measured in MRI. Comparison with brain pulse according to Schelten classification
leucoaraiosis load | one a year from inclusion visit to 5 years
  Measured in MRI. Comparison with brain pulse according to Fazekas classification
Carbohydrate metabolism | one a year from inclusion visit to 5 years
  Measured with PET-FDG in regions of interest involved in neurodegenerative diseases. Comparison with brain pulse
Spinal fluid biomarkers | one a year from inclusion visit to 5 years
  Determination of amyloid and tau proteins in spinal fluid. Comparison with brain pulse
cohort study on brain pulsatility with neuropsychological measures | one a year from inclusion visit to 5 years
  Comparison between brain pulsatility parameters and standard neuropsychological test scores used for cognitive assessment of patients with NCD.
  neuropsychological test scores are optional at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas DESMIDT, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided